CLINICAL TRIAL: NCT07172880
Title: Sedentary Behavior, Physical Activity, and 24-hour Behavior in Pregnancy and Offspring Health: the Pregnancy 24/7 Offspring Study
Brief Title: Pregnancy 24/7 Offspring Study
Status: Recruiting | Type: Observational
Sponsor: Kara Whitaker (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Pittsburgh (Other); West Virginia University (Other)
Responsible Party: Sponsor-Investigator, Kara Whitaker, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202211227; R01HL164662 (NIH)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Physical Activity; Sleep; Sedentary Behavior; Cardiovascular Disease Risk; Obesity Risk; Growth and Development; 24- Hour Movement Behaviors; Children; Pregnancy
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mother: Women who were enrolled in the Pregnancy 24/7 Cohort Study and subsequently delivered a live-born infant.
- Child: Children from birth to 30 months of age, born to participants enrolled in the Pregnancy 24/7 Cohort Study.

SUMMARY:
There is growing evidence that maternal health and behaviors in pregnancy, such as pre-pregnancy obesity, excessive gestational weight gain, poor diet, smoking, and adverse pregnancy outcomes, are linked to fetal programming for obesity and cardiovascular disease (CVD) risk in the offspring. Yet, there is a surprising lack of research on the role of prenatal sedentary behavior, physical activity, and sleep (conceptualized together as 24-hour behavior) on offspring obesity risk and CVD risk; this is an unfortunate research gap since there is strong physiological rationale that these behaviors in pregnancy could influence offspring health and are modifiable intervention targets in pregnancy. This multi-site observational cohort study will leverage state-of-the-art, 24-hour behavior assessment in each trimester of pregnancy, collected as part of the Pregnancy 24/7 cohort study and add additional assessments of offspring growth, adiposity, and CVD risk through 24 months to inform future primordial prevention interventions to decrease the risk of offspring obesity and CVD across the lifespan.

DETAILED DESCRIPTION:
Over the past three decades, there has been an alarming increase in the incidence of childhood obesity. Childhood obesity leads to early onset of cardiovascular risk factors, and both obesity and cardiovascular risk factors track into adulthood and contribute to the epidemic of cardiovascular disease (CVD). The Developmental Origins of Health and Disease theory posits that risk for obesity and CVD is, in part, programmed in utero. To prevent this early entrenchment into obesity and CVD, identification of modifiable maternal factors during pregnancy that later impact offspring risk in early childhood is essential. A surprising lack of research investigates the role of prenatal sedentary behavior (SED), moderate-to-vigorous-intensity physical activity (MVPA), and the novel 24-hour behavior paradigm (the composition of SED, physical activity, and sleep) on these adverse offspring outcomes. This is a critical research gap because there is strong physiological rationale that SED, MVPA, and 24-hour behavior in pregnancy could influence offspring health, and these behaviors are modifiable targets for intervention during pregnancy.

This project will address these research gaps with high rigor by leveraging the multi-center cohort study (Pregnancy 24/7, NCT04749849). In Pregnancy 24/7, SED, physical activity, and sleep were prospectively measured using state-of-the-art monitors (activPAL3 micro, Actiwatch Spectrum Plus), along with obesity, gestational weight gain, diet, smoking and adverse pregnancy and birth outcomes across pregnancy. In direct response to the NHLBI's NOT-HL-19-695, the scope of the Pregnancy 24/7 cohort study was expanded by conducting a separate cohort study in the participants' offspring (Pregnancy 24/7 Offspring Study). In the Offspring Study, maternal exposures (already collected in Pregnancy 24/7) will be combined with new, comprehensive assessments of the child's postnatal exposures and outcomes through 24 months. This approach will allow the investigative team to isolate the effects of pregnancy SED, MVPA, and 24-hr behavior on offspring growth and CVD risk measures in early childhood. Growth mixture modeling and state-of-the-art compositional data analyses will be used to address the following aims:

AIM 1: Examine associations of SED in pregnancy with offspring growth and CVD risk measures H1: Offspring of women with higher SED across pregnancy will have more rapid increases in BMIz (primary) and higher adiposity, blood pressure, and pulse wave velocity (secondary) through 24 months.

AIM 2: Examine associations of MVPA in pregnancy with offspring growth and CVD risk measures H2: Offspring of women with lower MVPA across pregnancy will have more rapid increases in BMIz (primary) and higher adiposity, blood pressure, and pulse wave velocity (secondary) through 24 months.

AIM 3: Determine optimal 24-hr behavior compositions in pregnancy to reduce the risk of adverse growth and CVD risk measures in the offspring H3: Statistically reallocating time in SED for LPA or MVPA, but not sleep (in adequate duration sleepers) across pregnancy will be associated with less rapid increases in BMIz (primary), and lower adiposity, blood pressure, and pulse wave velocity (secondary) in the offspring through 24 months.

By combining prenatal and postnatal exposure data, this approach uniquely allows the investigative team to isolate the effects of pregnancy SED, MVPA, and 24-hr behavior on offspring obesity and CVD risk measures in early childhood. This project will inform critically needed primordial prevention interventions to decrease the risk of obesity and CVD.

ELIGIBILITY:
Maternal Inclusion Criteria:

* Enrolled in Pregnancy 24/7 Study.
* Completed at least one 24-hr behavior assessment, with valid objective activity monitor data and questionnaires.
* Pregnancy resulted in singleton live birth.

Offspring Exclusion Criteria:

-Child diagnosed with congenital or chromosomal abnormalities that may affect growth or CVD risk.

Ages: 0 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women who participated in the Pregnancy 24/7 Cohort Study and gave birth who complete eligibility screening from three sites Iowa N=225, Pittsburgh N=112, and West Virgina N=113. We anticipate N=360 for 24-month chart abstraction and questionnaires and N=315 for the in-person visit, with approximately equal sex distribution among offspring.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-07-06 (Estimated); Study Completion 2027-07-06 (Estimated)

PRIMARY OUTCOMES:
BMIz | Through study completion for each participant: birth to 30 months old.
  BMI z-scores will be calculated using WHO growth standards from weight and length data abstracted from well-child visits (birth to 30 months; ~10 per child) and direct measurements at the 24-month study visit.

SECONDARY OUTCOMES:
Waist Circumference | 23-25 months old.
  Waist circumference will be measured at the 24- month study visit using a anthropometric tape to the nearest 1 mm.
Tricep and Subscapular Skinfolds | 23-25 months old.
  Subscapular and triceps skinfolds will be assessed at the 24- month visit in mm using a standard skinfold caliper on the right side of the body, with the mean value used. The sum of the mean values will be analyzed, along with WHO age- standardized z-scores for tricep and subscapular skinfolds.
Blood Pressure | 23-25 months old.
  Blood pressure will be assessed at the 24-month visit using a non-mercury aneroid sphygmomanometer following a 5-minute rest, with three readings taken at 1-minute rest intervals. The average of the second and third readings will be used.
Pulse Wave Velocity | 23-25 months old.
  Pulse wave velocity will be measured at the 24- month visit using the Vicorder® System, with cuffs placed on the upper arm and thigh inflated to 55 mmHg for 3-5 heart cycles. After a 5 minute rest, triplicate measurements will be completed in <5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Kara M Whitaker, PhD, MPH, Principal Investigator — University of Iowa; Bethany Barone Gibbs, PhD, Principal Investigator — West Virginia University; Sharon Ross, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified data that are relevant to the primary aims of the study will be made available along with a relevant data dictionary.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible, no later than the time of an associated publication, or the end of the award period, whichever comes first.
Access Criteria: Data access will be provided to external researchers who provide a methodologically sound proposal for secondary data analysis that is approved by the investigators of the study. Proposals should be directed to the study PI.